CLINICAL TRIAL: NCT02592915
Title: Monocentric, Prospective Randomized Controlled Clinical Trial Assessing the Effect on the Lower Limb Spinal Motoneuron Excitability, the Efficacy in Term of Morphinic Sparing and Safety of of Early Clonidine Bolus Intravenous Administration During General Anesthesia in Children and Adolescent 6-18 Years Old Requesting Reconstructive Tympanic Surgery
Brief Title: Effect of a Bolus of Clonidine Systemically Administered on the Excitability of the Spinal Motoneurons of the Lower Extremity
Acronym: EXCICLON
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: Brugmann University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: P2014/PE2
Record Dates: First submitted 2015-10-20; First posted 2015-10-30 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Intraoperative Neurophysiological Monitoring; Pain Management
MeSH Terms: conditions — Agnosia | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental): Patients randomized in the Test Group will receive the clonidine hydrochloride
  Interventions: Drug: Clonidine hydrochloride
- Control Group (Placebo Comparator): Patients randomized in the Control Group will receive the Placebo
  Interventions: Other: Single bolus of physiologic sodium chloride serum administered IV after induction and obtaining a stable anaesthetic level

INTERVENTIONS:
Drug: Clonidine hydrochloride — Single bolus of clonidine hydrochloride 0.3µg/kg (max 150 µg/kg) administered IV after induction and obtaining a stable anaesthetic level
  Arms: Test Group
Other: Single bolus of physiologic sodium chloride serum administered IV after induction and obtaining a stable anaesthetic level
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess the effect of IV clonidine administration on lower limb spinal motoneuron excitability during standardized total intravenous anesthesia (propofol and remifentanil).

DETAILED DESCRIPTION:
According to the literature data, intraoperative administration of clonidine reduces the need for morphine per and postoperative and thus reduces the side effects associated related to their administration.

Nevertheless, on the basis of current knowledge, clonidine may disrupt some electrophysiological measures required for the intraoperative monitoring of surgeries with a high risk of neurological complications.

For such surgery, anaesthesiologists are led to inject clonidine after surgery, at a time when the electrophysiological measures are no longer needed, which limits the benefit in terms of intraoperative morphine savings.

Whith this study, investigators would like to investigate if an early administration of clonidine in patients aged 6 to 16 years undergoing ear surgery disturbs excitability of the spinal motor neuron.

The choice of the study population is justified by the fact that the ear surgery does not require electrophysiological monitoring and it is carried out under conditions similar to that of anesthesia of scoliosis corrective surgery for which electrophysiological measurements are essential for the prevention of neurological complications.

Observations will allow investigators to determine therefore whether early administration of clonidine is possible at high risk of neurological complications surgeries for which electrophysiological monitoring is essential.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 6 to 18 years at time of hospital admission
2. Planned hospital admission for tympanoplasty
3. Informed Consent signed by both parents

Exclusion Criteria:

1. Known hypersensitivity to clonidine or to any component of the Catapressan
2. Patient treated with alpha2 agonists
3. Surgical emergency
4. Patient treated with antipsychotic drugs(butyrophenone, phenothiazine, tricyclic antidepressant)
5. Abnormal heart rhythms
6. Neuromuscular disease
7. Renal impairment
8. Patient treated with methylphenidate
9. Pregnant or breastfeeding woman

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the spinal motoneuron excitability through the measurement of the F wave before and after clonidine administration. | continuously during the surgery
Evaluation of the spinal motoneuron excitability through the measurement of H reflex before and after clonidine administration | continuously during the surgery

SECONDARY OUTCOMES:
Total dose of propofol and remifentanyl in mg/kg administered throughout the perioperative period | perioperative period, up to 5H
Pain score using the Children Hospital of Eastern Ontario Pain Scale (CHEOPS) or EVA scale | Every 30 minutes during the recovey period (up to 2H)
Sedative score using the University of Michigan Sedation Scale (UMSS) scale | Every 30 minutes during the recovery period (up to 2H)
Total dose of step 2 analgesic (tramadol) used for pain management | Total dose given during the recovery period (up to 2H)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Fabiola Children's University Hospital, Brussels, Belgium